CLINICAL TRIAL: NCT07113002
Title: EFFECTIVENESS OF EMOTIONAL FREEDOM TECHNIQUE FOR THE MANAGEMENT OF STRESS AND ANXIETY AMONG FEMALE HOSTELITES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Rija Munir, Principal Investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJWU/EC/2024/80
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Stress and Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (EFT) (Experimental): Participants received 4 weeks of Emotional Freedom Technique (EFT) therapy.
  Interventions: Behavioral: Emotional Freedom Technique (EFT)
- Control Group (No Intervention): Participants in this group did not receive Emotional Freedom Technique (EFT) therapy. They served as the control group for comparison with the intervention group.

INTERVENTIONS:
Behavioral: Emotional Freedom Technique (EFT) — Emotional Freedom Technique (EFT) is a psychological intervention that uses tapping on acupuncture points combined with cognitive techniques to reduce stress and anxiety. Participants received EFT sessions for 4 weeks.
  Arms: Intervention Group (EFT)

SUMMARY:
This study tested how well Emotional Freedom Technique (EFT) works to reduce stress and anxiety in female university students living in hostels. Eighty students were randomly divided into two groups: one received EFT therapy for 4 weeks, and the other did not. Stress and anxiety were measured before and after using standard scales. The group that received EFT showed a significant reduction in stress and anxiety compared to the control group. This suggests EFT is an effective way to help manage mental health problems in this group.

ELIGIBILITY:
Inclusion Criteria:

* Female students living in university hostels.

Female students who have provided informed consent to participate.

Exclusion Criteria:

* Male students.

Hostel professionals and management living in hostels.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligible participants are self-identified females only.
Enrollment: 80 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
Reduction in Stress Levels | Baseline and 4 weeks after intervention
  Stress levels measured using the Perceived Stress Scale (PSS-10) to assess the effect of Emotional Freedom Technique (EFT) therapy on stress reduction among female hostelites.

SECONDARY OUTCOMES:
Reduction in Anxiety Levels | Baseline and 4 weeks after intervention
  Anxiety levels measured using the Generalized Anxiety Disorder scale (GAD-7) to evaluate the effect of Emotional Freedom Technique (EFT) therapy on anxiety reduction among female hostelites.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Rayan Hostel, Rawalpindi, Punjab Province, Pakistan